CLINICAL TRIAL: NCT01858909
Title: Phase III, Prospective, Randomized, Double-blind Clinical Trial to Evaluate the Efficacy of Melatonin in Patients With Severe Sepsis or Septic Shock
Brief Title: Efficacy of Melatonin in Patients With Severe Sepsis or Septic Shock
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aragon Institute of Health Sciences (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRA-172
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Melatonin; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): saline every 12 hours for 28 days
- Melatonin (Experimental): Oral 30mg/12hours melatonin 28 days
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Administration via oral or via a nasogastric tube followed by 20mL saline
  Other Names: Liquid 1 mg/mL Melatonin
  Arms: Melatonin

SUMMARY:
OBJECTIVES. To establish the therapeutic efficiency of melatonin in adult patients with severe sepsis and septic shock.

Specifically:

1. To evaluate the survival to 28 days of mechanical assisted ventilation, days with vasoactive drugs, need of hemodialysis-hemofiltration, superinfection and evolution towards the failure of other organs.
2. To evaluate, waiting for reduction under the influence of the treatment with melatonin, :

   1. clinical - analytical parameters of sepsis;
   2. levels of cytokines;
   3. oxidative and nitrosative stress;
   4. acute-phase proteins (APP), specially of the ITIH4;
   5. immune response;
   6. endocrine response.

METHODOLOGY. Patients will be randomized in two groups, n = 55 in each group: 1) treatment with melatonin 30mg/12 hours 28 days; 2) placebo.

Determinations: a) clinical - analytical parameters relative to the sepsis; b) melatonin plasmatic levels; c) quantification of malonyldialdehyde and 4-hydroxynonenal, protein carbonyl content, nitrites, erythrocyte membrane fluidity, and superoxide dismutase, catalase, glutathione reductase and glutathione peroxidase activity; d) Interleukins-1,2,4,5, 6, 7,8,10,12,13, IFN-γ; TNF-α and GM-CSF; e) acute-phase proteins: PCR, haptoglobin, Apo A-I, α1-GPA and ITIH4; f) lymphocytes T, B, NK, T CD4, and T CD8, and immunoglobulins; g) cortisol, aldosterone, ACTH, ADH, insulin, glucagon and 25-hydroxyvitamin D3. Data will be analyzed following a prospectively define plan and by intention-to-treat (ITT) analysis.

DETAILED DESCRIPTION:
This study will be done in the Hospital Clinico Lozano Blesa (Zaragoza, Spain), promoted by the Health Science Aragon Institute and its principal investigator is F. Agustín García Gil (Surgical Service). It will start in April-May 2013 and will finish 12 months later approximately. The study sponsor is I+CS (Aragon Institute of Health Sciences).

ELIGIBILITY:
Inclusion Criteria:

* patients (males and females) over 18 years who meet the diagnostic criteria for severe sepsis or septic shock secondary to community-acquired pneumonia or hospital and or intra-abdominal infection

Exclusion Criteria:

* Patient with more than 24 hours from the first documentation of organ dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 month
  Mortality at 28 days of study entry.
Clinical evolution parameters | 1 month
  Days of mechanical ventilation. Days with vasoactive drugs. Days with hemodialysis or hemofiltration. Superinfection of organs other than the initial cause of the sepsis. Progression to other organs fail after starting the treatment.

SECONDARY OUTCOMES:
Clinical evolution | 1 month
  clinical - analytical parameters relative to the sepsis
Oxidative-nitrosative parameters | 1 month
  Melatonin plasmatic levels Quantification of malonyldialdehyde and 4-hydroxynonenal Protein carbonyl content Nitrites Erythrocyte membrane fluidity Superoxide dismutase, catalase, glutathione reductase and glutathione peroxidase activity
Inflammatory parameters | 1 month
  Interleukins-1,2,4,5, 6, 7,8,10,12,13, IFN-γ; TNF-α and GM-CSF
Acute phase proteins | 1 month
  PCR, haptoglobin, Apo A-I, α1-GPA and ITIH4
Immune parameters | 1 month
  Lymphocytes T, B, NK, T CD4, and T CD8, and immunoglobulins
Endocrine parameters | 1 month
  Cortisol, aldosterone, ACTH, ADH, insulin, glucagon and 25-hydroxyvitamin D3

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A García-Gil, Physician, Principal Investigator — Hospital Clínico Universitario Lozano Blesa
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza, Spain